CLINICAL TRIAL: NCT04904562
Title: Angiotensin II as a First-line Vasopressor for Distributive Shock During or After Heart Transplantation or Durable Left Ventricular Assist Device Implantation: A Pilot Study
Brief Title: Angiotensin II for Distributive Shock
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Northwestern University (Other)
Collaborators: La Jolla Pharmaceutical Company (Industry)
Responsible Party: Principal Investigator, Choy Lewis, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: STU00211528
Record Dates: First submitted 2021-05-12; First posted 2021-05-27 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Distributive Shock
Keywords: Vasoplegia
MeSH Terms: conditions — Vasoplegia | interventions — Angiotensin II; Giapreza; Saline Solution

STUDY DESIGN:
Intervention Model Description: 1:1 randomization to receive either study drug or placebo
Who Masked: Participant, Care Provider, Investigator
Masking Description: Study medication and matching placebo (saline) administered by IV infusion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Active Comparator): Angiotensin II administered as an intravenous (IV) infusion will be increased every 5 minutes by 5-10ng/kg/min increments up to 80ng/kg/min
  Interventions: Drug: Angiotensin II
- Control (Placebo Comparator): Intravenous (IV) infusion (saline)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Angiotensin II — Angiotensin II started at 5 ng/kg/min and titrated in 5-10 ng/kg/min increments every 5 minutes up to 80ng/kg/min to achieve target arterial pressure (MAP)
  Other Names: Giapreza
  Arms: Treatment
Drug: Placebo — Placebo
  Other Names: Saline solution
  Arms: Control

SUMMARY:
This is a single-center, randomized, double-blind, placebo-controlled pilot study. A total of 40 patients who develop distributive shock, intra-operatively or post-operatively within 48 hours of heart transplant or left ventricular assist device placement will be enrolled. Participants will be randomized to Angiotensin II (Giapreza) vs. placebo plus standard of care, as a first line agent for vasoplegia. Two groups of patients will be enrolled:

* Group A: Heart Transplant (10 control, 10 treatment)
* Group B: LVAD implant (10 control, 10 treatment)

DETAILED DESCRIPTION:
Patients undergoing implantation of a durable left ventricular assist devices (LVAD) or a heart transplantation are at increased risk for cardiac vasoplegia. Vasoplegia, during or following cardiac surgery, is a life-threatening condition that is characterized by poor organ perfusion and may progress to multi-organ failure. The prognosis is especially poor for patients with refractory hypotension, despite high doses of vasopressors. Existing data point to total catecholamine dose, cumulative time spent with hypotension, volume overload, need for blood transfusion as contributing factors. Catecholamine vasopressors and vasopressin, which are often used as first line vasopressor therapy, are also independent risk factors for end organ dysfunction. Data comparing mortality with the use of different classes of vasopressors, in various types of shock, have been equivocal to date. In addition, data comparing the use of different classes of vasopressors for vasoplegia during or after heart transplantation and LVAD implantation are lacking. In patients with distributive shock in the intensive care unit, angiotensin II has been shown to reduce total catecholamine dose over 24 hours and the cumulative time spent with hypotension. This study will evaluate, as the primary endpoint, whether first line use of angiotensin II affects total catecholamine vasopressor dose in the first 24 hours after vasoplegia is first. Secondary endpoints include cumulative time spent with mean arterial pressure < 70 mmHg within the first 24 hours after distributive shock is first diagnosed, need for vasoplegia rescue therapies (methylene blue, vitamin B12, Vitamin C, steroids), incidence of acute kidney injury and stroke, time to extubation, incidence of new tachyarrhythmias, need for blood transfusion and fluid overload within the first 24 hours, ICU and hospital length of stay, 30-day mortality and allograft rejection (for heart transplant recipients).

ELIGIBILITY:
Inclusion Criteria:

1. Patients (18 years of age or older)
2. Onset of distributive shock within 48 hours after heart transplantation or VAD placement. Distributive shock defined as MAP less than 55mmHg on CPB, MAP less than 70mmHg before or after CPB, or systemic vascular resistance (SVR) less than 800 dynes/cm/sec5 with cardiac index (CI) greater than 2.0L/min/m2 and clinically determined euvolemia.

Exclusion Criteria:

1. Patients without distributive shock,
2. Women who are pregnant or breastfeeding.
3. Patients who do not receive the study drug as a first line agent for distributive shock
4. Allergy to angiotensin II, angiotensin II or another vasopressor being used at the time of presentation to the operating room
5. Preexisting distributive shock
6. Preexisting thromboembolic disease
7. Patients who are unwilling to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Total catecholamine dose | 24 hours
  Total catecholamine dose for first 24 hours after distributive shock is first diagnosed

SECONDARY OUTCOMES:
Cumulative time spent with MAP < 70 mmHg | 24 hours
  Cumulative time spent with MAP < 70 mmHg within the first 24 hours after distributive shock is first diagnosed
Time to extubation | 24 hours
  Time to extubation after arrival in the ICU if distributive shock is diagnosed intraoperatively or time to extubation after distributive shock is diagnosed postoperatively
Incidence of stroke | 48 hours
  Incidence of stroke confirmed by neurologist within 48 hours after distributive shock is first diagnosed
Incidence of acute kidney injury | 48 hours
  Incidence of acute kidney injury, staged by KDIGO Creatinine criteria, within 48 hours after distributive shock is first diagnosed
Incidence of new tachyarrhythmia | 24 hours
  Incidence of new tachyarrhythmia within the first 24 hours after distributive shock is first diagnosed
Units of blood transfused | 24 hours
  Units of blood transfused within first 24 hours after distributive shock is first diagnosed
Fluid overload | 24 hours
  Fluid overload within the first 24 hours after distributive shock is first diagnosed
Intensive care unit (ICU) length of stay | 1 year
  Total time spent in the ICU after initial diagnosis of distributive shock
Hospital length of stay | 1 year
  Total time spent in the hospital after diagnosis of distributive shock
30-day mortality | 30 days
  Subject death within 30 days of diagnosis of distributive shock

CONTACTS AND LOCATIONS:
Overall Officials: Choy Lewis, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided